CLINICAL TRIAL: NCT06492447
Title: Correlation Study of Serum HER 2 Against HER 2-ADC Drug Efficacy in HER 2 Low-expressing Breast Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Shenzhen New Industries Biomedical Engineering Co., Ltd. (Unknown)
Responsible Party: Sponsor
Other Study IDs: HR-BLTN-016
Record Dates: First submitted 2024-07-02; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: HER 2 Low-expressing Breast Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HER2 low-expressing
  Interventions: Drug: Against HER 2-ADC Drug

INTERVENTIONS:
Drug: Against HER 2-ADC Drug — Breast cancer subjects receiving anti-HER2-ADC drugs were treated with a 3-week treatment cycle lasting 6 cycles. Serum of patients before and after treatment was collected, and the changes of serum HER2 level before chemotherapy and after 2, 4 and 6 cycles of chemotherapy were dynamically monitored, and the relationship between HER2 level and the therapeutic effect of different targeted drugs was analyzed.

SUMMARY:
Breast cancer is one of the most common malignancies in women worldwide, with HER2-positive breast cancer accounting for about 15-20% of all breast cancer cases. HER2 (Human epidermal growth factor receptor 2) is a tyrosine kinase receptor that, when overexpressed, promotes the growth and spread of tumor cells. The advent of anti-HER2 therapy, particularly antibody-coupled drugs (ADCs), has resulted in significant survival benefits for HER2-positive breast cancer subjects.

At present, the value of serum HER2 in the monitoring of anti-HER2-ADC drug therapy is insufficient. The purpose of this study was to investigate changes in serum HER2 expression levels in breast cancer subjects treated with anti-HER2-ADC drugs and the relationship between these changes and treatment effect. The therapeutic effect of HER2 was evaluated by continuous detection of HER2 serum, which provided a theoretical basis for the selection of clinical drug treatment.

DETAILED DESCRIPTION:
ADC drugs are a new type of targeted therapy. ADC drugs are composed of monoclonal antibodies, linkers and drug carriers, which bind to the target antigen on the surface of tumor cells through antibodies, endocytosis/internalization to form early endosomes in cells, and then mature into late endosomes and fuse with lysosomes. ADC drugs break apart in the lysosome and release the drug carrier, eventually leading to apoptosis or death while minimizing damage to normal cells. However, not all subjects with HER2-positive breast cancer respond well to ADC drugs, and resistance may develop during treatment. Therefore, effective biomarkers are needed to monitor treatment effects and guide individualized treatment. Serum HER2 refers to the HER2 protein fragment present in the subject's serum. Serum HER2 levels may be more readily available than HER2 expression in tumor tissue and can be sampled multiple times during treatment, allowing real-time monitoring of disease progression and drug efficacy. If monitoring of serum HER2 levels accurately reflects tumor sensitivity to ADC drugs, it could be a valuable therapeutic monitoring tool.

In view of the excellent efficacy of ADC drugs in HER2-positive and low-expression breast cancer patients, this study intends to judge the therapeutic efficacy of breast cancer patients treated by anti-HER2-ADC drugs (such as T-DXd) through continuous detection of their serum HER2, providing a theoretical basis for the selection of clinical drug therapy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects with pathologically confirmed breast cancer; 2. The therapeutic drugs are anti-HER2-ADC drugs; 3. No history of other tumors; 4. Age > 18 years old; 5. Have relatively complete clinical case characteristics data.

Exclusion Criteria:

* 1. Male breast cancer subjects; 2. Suffering from other malignant neoplasms; 3. Subjects with incomplete clinical case characteristics.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients treated with anti-HER2-ADC drugs
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-07-04 (Estimated); Primary Completion 2026-01-04 (Estimated); Study Completion 2026-03-04 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 1-2 years
  Percentage of patient's measurable disease who have achieved either complete response (CR) or partial response (PR) according to RECIST 1.1.

SECONDARY OUTCOMES:
PFS | 1-2 years

IPD SHARING:
Plan to Share IPD: Undecided